CLINICAL TRIAL: NCT01871870
Title: Sensor-controlled Insulin- and Glucagon Delivery in Subjects With Type 1 Diabetes: Testing of an Automated System in an Outpatient (Hotel) Setting.
Brief Title: Artificial Pancreas Control System in an Outpatient Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013.001
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artificial Pancreas Control Software (Experimental): Type 1 Diabetes Mellitus subjects who fit the inclusion/exclusion criteria will undergo artificial pancreas closed-loop study for 28 hours. For the entire study, the adaptive component of Artificial Pancreas Control Software will be used to control the subject's blood glucose.
  Interventions: Device: Artificial Pancreas Control Software

INTERVENTIONS:
Device: Artificial Pancreas Control Software — This master controller software is used in conjunction with two subcutaneous continuous glucose monitoring systems and two Omnipod pumps, one for administering aspart insulin (NovoLog) and one for administering glucagon (GlucaGen), to control blood glucose levels. The insulin and glucagon infusion rates are determined by an outpatient automated version of the Adaptive Proportional Derivative (APD) insulin and glucagon control algorithm programmed into a smart phone.

SUMMARY:
The objectives of this outpatient research study are (1) to assess the ability of this automated system to be operated by a subject with limited professional oversight; (2) to assess whether the new devices (Dexcom Gen 4 sensors, Motorola ES400 smart phone, iDex pump controller) will reduce the frequency of hardware and data communication lapses seen in the previous system; and (3) to measure the degree of glucose control achievable with this automated system. The system will adjust blood glucose by administering insulin and glucagon. Insulin is a hormone that lowers blood glucose and will be given nearly continuously during this study. Glucagon raises blood glucose and will be automatically administered during hypoglycemia. Both are natural hormones made by people without diabetes. Each subject will have four devices placed on his abdomen: two Omnipod insulin pumps, one for delivering insulin and one for delivering glucagon, and two Dexcom G4 glucose sensors for measuring glucose. The two sensors will feed glucose data into Motorola smart phone master controller, which will calculate the correct amount of insulin or glucagon to deliver. The system will then send the command to the correct Omnipod through the iDex pod controller.

In this new system, the research subject will be able to monitor the progress of the study by use of the smart phone graphical user interface. The subject will have a companion with him/her during the entire study for safety purposes. Both the subject and companion will complete a training course on how to treat diabetic emergencies and how to operate the system. A study physician and technician will be in the hotel during each study and will be monitoring the study via a cloud-based data communication system. These studies will be carried out in a hotel setting.

DETAILED DESCRIPTION:
The objective of the current human study is to verify the components of the Artificial Pancreas Control Software during an outpatient study. This master controller software is designed to be used in conjunction with two subcutaneous continuous glucose monitoring systems to regulate blood glucose levels as well as two Omnipod pumps, one for administering insulin and one for administering glucagon. The sensors communicate wirelessly with two sensor receivers which will be interfaced with the APC by wireless USB connection. The insulin and glucagon pumps will be controlled by the APC through a wireless USB connection. The algorithm included in the APC is an automated version of the Adaptive Proportional Derivative (APD) insulin and glucagon control algorithm, which was previously studied as an investigational device. The Automated APD has been studied in vivo (in 13 experiments, each 28 hr in length, with automated adjustment of pumps) and no serious adverse effects were noted. The APC will be tested in vivo during 28 hour experiments in an outpatient setting in preparation for home testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 21 to 60 years of age.
* Current use of an insulin pump.
* Willingness to follow all study procedures and to stay with a companion during the outpatient test of the artificial pancreas.
* Willingness to sign informed consent and HIPAA documents.
* Willingness for the subject and companion to attend a training course on the system including emergency management of extremes of glucose.

Exclusion Criteria:

* Pregnancy or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Renal insufficiency (serum creatinine of 2.0 mg/dL or greater).
* Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less than 3.3 g/dL; or serum bilirubin of over 2.
* Adrenal insufficiency
* Hematocrit of less than or equal to 34%.
* A history of cerebrovascular disease or coronary artery disease regardless of the time since occurrence.
* Congestive heart failure, NYHA class III or IV.
* Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Any active infection.
* Visual impairment preventing reading of glucose meter values or continuous glucose monitoring device.
* Physical impairment impeding the ability to use a glucose meter or continuous glucose monitoring device.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator).
* Active malignancy, except basal cell or squamous cell skin cancers.
* Major surgical operation within 30 days prior to screening.
* Seizure disorder even if controlled by stable therapeutic regimen.
* Current administration of any beta blocker medication, clonidine, reserpine, or guanethidine
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Current administration of oral or parenteral corticosteroids.
* Use of an investigational drug within 30 days prior to screening.
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Allergy to glucagon.
* Past history of pheochromocytoma or a family history of MEN 2, neurofibromatosis, or von Hippel-Lindau disease.
* Insulin resistance requiring more than 200 units per day.
* Need for uninterrupted treatment of acetaminophen.
* History of hypoglycemic unawareness.
* C peptide level of ≥0.5 ng/ml
* Any reason the principal investigator deems exclusionary.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K Ward, MD, Principal Investigator — Legacy Health
Locations (1):
- Legacy Research Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Artificial Pancreas Control Software
Started | 20
Completed | 11
Not Completed | 9
Not completed — Hardware issues | 7
Not completed — hyperglycemia | 2

BASELINE CHARACTERISTICS:
Arm/Group | Artificial Pancreas Control Software
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Verification of the Automation and Telemetry Components
Description: This outcome will verify afferent signal transmittal from the Dexcom sensors to the algorithm and the efferent signal transmittal from the algorithm to the insulin and glucagon pumps. Outcome measure is the average number of sensor and/or pump telemetry failures per 28 hour study.
Time Frame: 28 hours
Measure: Mean (Standard Deviation); unit: failures
Arm/Group | Artificial Pancreas Control Software
Number analyzed (Participants) | 20
failures | 16.5 (8)

2. Secondary Outcome: Deviation From Target Blood Glucose
Description: Assessment of how accurately the algorithm controls glycemia in the subjects will be carried out using the mean deviation from the target blood glucose (mg/dL). Deviation is measured as algorithm controlled glucose level minus target glucose level.
Time Frame: 28 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Artificial Pancreas Control Software
Number analyzed (Participants) | 20
mg/dl | 91.35 (91.41)

ADVERSE EVENTS:
Arm/Group | Artificial Pancreas Control Software
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas Control Software (N=20)
nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes